CLINICAL TRIAL: NCT04694287
Title: Volume Flow Assessment to Optimize Angioplasty of Dysfunctional Dialysis Access. The VOLA II Multicenter Study
Brief Title: Volume Flow Assessment to Optimize Angioplasty of Dysfunctional Dialysis Access
Acronym: VOLAII
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Collaborators: University Hospital of Patras (Other); Nefrolgiki SA Hemodialysis Center (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Associate Professor of Interventional Radiology, Attikon Hospital
Other Study IDs: EBD 692
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Dialysis Access Malfunction
Keywords: Percutaneous transluminal angioplasty; Volume-flow measurement; Autologous arteriovenous fistula; Dialysis access; Interventional Radiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volume flow group: The study will include consecutive patients undergoing standard fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF. Intraprocedural volume flow measurements will be obtained just prior to the procedure and after final balloon dilation.
  Interventions: Diagnostic Test: Percutaneous DUS volume flow measurements

INTERVENTIONS:
Diagnostic Test: Percutaneous DUS volume flow measurements — Volume flow measurements of the AFV will be obtained using intraprocedural DUS just prior to sheath insertion and at the end of the final balloon dilation, before sheath removal.

SUMMARY:
This is a multicenter, prospective study investigating a new concept of intra-procedural percutaneous duplex ultrasound (DUS) volume flow-guided balloon angioplasty for the quantification and optimization of endovascular treatment outcomes of dysfunctional autologous arteriovenous fistulae (AVF).

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm observational clinical trial investigating a new functional index of success of endovascular treatment of dysfunctional AVF assessed with intraprocedural percutaneous DUS. The study will include 100 consecutive patients undergoing fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF. Exclusion criteria will be (i) patients with arteriovenous synthetic grafts. (ii) Immature AFVs not previously used for hemodialysis (at least once). Patients' demographical data, dialysis access history, and procedural details will be recorded. Intraprocedural volume flow measurements will be obtained just prior to the procedure and after final balloon dilation, before sheath removal. Clinical follow-up will be set at 6 months after the index procedure. All DUS measurements will be performed using the same imaging protocol. The study's primary endpoints will be (i) the quantification of angioplasty outcome using DUS volume flow analysis before sheath insertion and at the end of the procedure before sheath removal and (ii) to assess the correlation between volume flow at the end of the procedure and clinically driven re-intervention-free rate at defined as the rate of reintervention due to dysfunction recurrence of the treated AVF. Secondary endpoints will be (i) to assess the correlation between volume flow and clinical success defined as high-quality dialysis for a period of at least one month and (ii) identification of independent predictors of re-intervention-free rate.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF
* Signed consent form
* Agree to the study protocol

Exclusion Criteria:

* Patients with arteriovenous synthetic grafts
* Patients with contraindication to antiplatelet therapy
* Immature AFVs, not previously used for at least one dialysis session.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing fluoroscopically-guided percutaneous balloon angioplasty due to dysfunctional AVF and assessed with pre-and post-procedural volume flow measurements using percutaneous DUS
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Quantification of angioplasty outcome | At the end of the procedure
  The quantification of angioplasty outcomes will be performed using DUS volume flow analysis
Correlation between volume flow and clinically-driven reintervention rate | 6 months
  The investigators will use ROC analysis to define cut off values of volume flow at the end of the procedure to predict clinically-driven reintervention rate

SECONDARY OUTCOMES:
Re-intervention-free rate | 6 months
  The clinically driven re-intervention-free rate due to dysfunction recurrence of the treated AVF following endovascular treatment
Identification of independent predictors of reintervention | 6 months
  Multivariable analysis will be performed to identify independent predictors of reintervention-free rate
Procedure related complications | 1 week
  Minor and major procedure related complications will be recorded

CONTACTS AND LOCATIONS:
Locations (3):
- Greece (3):
  - Patras Universityu Hospital, Pátrai, Achaia
  - "Attikon" University General Hospital, Athens, Attica
  - Nefrologiki SA Hemodialysis Centre, Athens, Attica

IPD SHARING:
Plan to Share IPD: Yes
Available after study publication, upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 1 month after publication and for 2 years
Access Criteria: Reasonable request (systematic review, metaanalysis)

REFERENCES:
- [Derived] Spiliopoulos S, Filippou P, Giannikouris IE, Katsanos K, Palialexis K, Grigoriadis S, Kitrou P, Brountzos E, Karnabatidis D. US Volume Flow Assessment to Optimize Angioplasty of Dysfunctional Dialysis Access: The VOLA-II Multicenter Study. Radiology. 2024 Nov;313(2):e233076. doi: 10.1148/radiol.233076. PMID 39589250